CLINICAL TRIAL: NCT01876329
Title: Presence of Autoantibodies to Gastric Parietal Cells and Subsequent Vitamin B12 Deficiency in Rheumatoid Arthritis Patients
Brief Title: Autoantibodies to Gastric Parietal Cells in Rheumatoid Arthritis Patients
Status: Completed | Type: Observational
Sponsor: Keesler Air Force Base Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Matthew B. Carroll, LtCol, USAF, MC, FACP, FACR, Chief of Rheumatology, Keesler Air Force Base Medical Center
Other Study IDs: FKE20130010H
Record Dates: First submitted 2013-06-09; First posted 2013-06-12 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Vitamin B12 Deficiency
Keywords: Rheumatoid Arthritis; Vitamin B12 deficiency; Autoimmune Thyroid Disease; Autoantibodies
MeSH Terms: conditions — Vitamin B 12 Deficiency; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Rheumatoid Arthritis: Patients with seropositive or seronegative Rheumatoid Arthritis
- Autoimmune Thyroid Disease (AITD): Participants with autoimmune thyroid disease without other known systemic or organ specific autoimmune illnesses.
- Control: Participants without Rheumatoid Arthritis, AITD, or other systemic or organ specific autoimmune illnesses

SUMMARY:
A review of the literature reveals that very few studies have assessed the potential co-existence of vitamin B12 deficiency due to gastric parietal cell autoantibodies. While Segal et al. in 2004 published a study which found that 49% of patients with RA had vitamin B12 deficiency, no assessment of the etiology or the presence of autoantibodies was made. While Goeldner et al. in 2011 and Datta et al. in 1990 demonstrated that anti-gastric parietal cell antibodies (anti-GPC Ab) were found in <5% to 28% of RA patients respectively, no additional testing was implemented to determine the significance, specifically whether or not the presence of anti-GPC Ab related to vitamin B12 deficiency.

The purpose of this study is to determine the prevalence and metabolic significance of anti-GPC Ab in three cohorts: (1) a group of patients with Rheumatoid Arthritis, (2) a group of patients with autoimmune thyroid disease (AITD), and (3) a group of patients with neither RA or AITD. To determine the significance of the presence of anti-GPC Ab, testing of the current serum B12 level along with a metabolite dependent on adequate vitamin B12 levels (Methylmalonic acid) will be tested.

DETAILED DESCRIPTION:
Background: Organ specific antibodies such as anti-gastric parietal cell antibodies (anti-GPC Ab) have been found in a variable number of patients with RA, but it is unclear what significance these antibodies have on actual vitamin B12 levels. Patients with RA have been found to have vitamin B12 deficiency up to near 50% but it is unclear if this deficiency is due to anti-GPC Ab.

Hypothesis: By virtue of the aberrant autoimmune process that occurs in RA, patients with RA are more likely to have anti-GPC Ab and more likely than a control arm or participants with autoimmune thyroid disease (AITD) to have vitamin B12 deficiency.

Method: 135 patients will be consented; 45 to the RA arm, 45 to an AITD arm, and 45 to a control arm. Exclusion criteria will filter patients who would have other reasons for altered vitamin B12 absorption, such as inflammatory bowel disease, surgery, or medication use. After obtaining consent subjects will be sent to lab a serum anti-GPC Ab test (obtainable in an SLE panel), RF, B12/folate (as available for ordering in CHCS), methyl malonic acid, and (for the control arm subjects and AITD subjects) an anti-CCP IgG. Patients will also complete a one-sided, one page questionnaire asking them about dietary and medication exposures.

Outcomes: (1) Determine whether evidence of serum vitamin B12 deficiency, as measure by either a low vitamin B12 level or elevated methylmalonic acid, will be more common in RA patients with anti-GPC Ab. (2) Determine the prevalence of anti-GPC Ab in a group of patients with RA as compared to a group of patients with AITD and with no known systemic or organ specific autoimmune condition.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age 18 and older
* RA arm: History of Rheumatoid Arthritis
* AITD arm: History of an autoimmune thyroid disease without a history or clinically obvious manifestation of an organ specific or systemic autoimmune process.
* Control arm: No history of RA and no history or clinically obvious manifestation of an organ specific or systemic autoimmune process.

Exclusion Criteria:

* Known vitamin B12 deficiency for which the participant was formerly treated or continues to receive therapy.
* Active malabsorptive state to include but not limited to celiac disease, inflammatory bowel disease, etc.
* Surgically induced malabsorptive state to include but not limited to Roux-en-Y Gastric bypass
* Use of medications that may interfere with vitamin B12 absorption
* Patients with a thyroid condition not consistent with an autoantibody process (i.e. congenital absence of the thyroid, infectious thyroiditis, thyroidectomy for non-autoimmune process, toxic multinodular goiter) will be excluded from the autoimmune thyroid arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Internal Medicine and Internal Medicine Specialty Clinics at one academic community hospital.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2013-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Carroll, MD, Principal Investigator — Keesler Medical Center
Locations (1):
- Keesler Medical Center, Keesler Air Force Base, Mississippi, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rheumatoid Arthritis | Autoimmune Thyroid Disease (AITD) | Control
Started | 45 | 36 | 44
Completed | 45 | 36 | 44
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rheumatoid Arthritis | Autoimmune Thyroid Disease (AITD) | Control | Total
Number analyzed (Participants) | 45 | 36 | 44 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 32 | 25 | 33 | 90
  >=65 years | 13 | 11 | 11 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (13.1) | 55.1 (17.2) | 55.8 (16.4) | 56.8 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 31 | 95
  Male | 11 | 6 | 13 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 10 | 3 | 7 | 20
  White | 33 | 28 | 34 | 95
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Vitamin B12 Deficiency
Description: Hypothesis: Evidence of serum vitamin B12 deficiency, as measure by either a low vitamin B12 level or elevated methylmalonic acid, will be more common in RA patients with anti-GPC Ab.
Time Frame: 7 months
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis | Autoimmune Thyroid Disease (AITD) | Control
Number analyzed (Participants) | 45 | 36 | 44
participants | 3 | 6 | 4

2. Secondary Outcome: Presence of Anti-GPC Antibodies
Description: Hypothesis: Evidence of anti-GPC Ab in a group of patients with RA will be more prevalent as compared to a group of patients with AITD and with no known systemic or organ specific autoimmune condition.
Time Frame: 7 months
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis | Autoimmune Thyroid Disease (AITD) | Control
Number analyzed (Participants) | 45 | 36 | 44
participants | 7 | 4 | 8

ADVERSE EVENTS:
Arm/Group | Rheumatoid Arthritis | Autoimmune Thyroid Disease (AITD) | Control
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/36 | 0/44
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes